CLINICAL TRIAL: NCT04061031
Title: Improving Self-Regulation Among Adopted Children: A Randomized Controlled Feasibility Trial
Brief Title: Improving Self-Regulation Among Adopted Children
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Brian Allen, Associate Professor, Department of Psychiatry, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12662
Record Dates: First submitted 2019-08-16; First posted 2019-08-19 (Actual); Last update posted 2021-12-16 (Actual); Status verified 2021-12

CONDITIONS: Self-regulation
Keywords: Self-regulation, adoption, parent-child realtionship
MeSH Terms: conditions — Self-Control

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Parent-Child Interaction Therapy (Experimental)
  Interventions: Behavioral: Parent-Child Interaction Therapy (PCIT)
- Child-Centered Therapy with Parent Education (Active Comparator)
  Interventions: Behavioral: Child-Centered Therapy with Parent Education

INTERVENTIONS:
Behavioral: Parent-Child Interaction Therapy (PCIT) — A trained clinician teaches the caregiver to deliver a number of behavior modification techniques for use with the child and coaches the caregiver in the delivery of those techniques.
  Arms: Parent-Child Interaction Therapy
Behavioral: Child-Centered Therapy with Parent Education — A trained clinician delivers non-directive, child-centered treatment techniques with the child while providing education to the parent based on current recommendations from the Department of Health and Human Services' Child Welfare Information Gateway.
  Other Names: Treatment-as-Usual
  Arms: Child-Centered Therapy with Parent Education

SUMMARY:
The proposed study will examine two different intervention programs and whether they improve self-regulation of adopted children. The study is a small randomized controlled trial to test the feasibility of conducting a larger, R01-funded clinical trial. Outcomes will primarily be focused on feasibility concerns, such as recruitment and retention of a sufficient number of participants and implementation of treatment protocols with fidelity, as well as determining initial effect size estimates that might inform later power analyses and examining the functioning of developmental assessment measures when administered in the context of a clinical trial.

DETAILED DESCRIPTION:
In the year 2016, over 57,000 children were adopted from the child welfare system and another 118,000 were awaiting adoption, an increase of 7.9% and 8.1%, respectively, since 2013. Children adopted from the child welfare system, on average, display significant and often profound challenges with self-regulation, defined as the external and internal processes responsible for determining one's emotional, behavioral, and cognitive reactions to stimuli. Poor self-regulation is linked to a host of later untoward outcomes. Permanency for children through the process of adoption offers an opportunity for improving developmental trajectories and later outcomes for children. Psychosocial interventions that can significantly improve the parent-child relationship hold promise for increasing the success of the adoption and further promoting healthy development for children. Prior to proceeding with an R01 application and funded clinical trial, a feasibility study is required for multiple reasons. First, it is necessary to determine the likelihood of recruiting and retaining a sufficient number of participants, the extent to which participants attend sessions on a regular basis, caregiver satisfaction with treatment, and potential barriers to clinicians implementing the intervention protocols with fidelity (Specific Aim 1), Second, a number of developmental measures will be implemented to examine improvement. These measures are typically administered in longitudinal developmental research, not clinical research, and the sensitivity of these tools to change is unknown. Therefore, this project will allow for a pilot examination of the implementation of these tools in a clinical context and the extent to which change may occur (Specific Aim 2). Finally, effect size estimates of change for key outcome metrics (i.e., self-regulation, parent-child relationship) will be derived to inform power analyses and sample size determinations for an R01 application (Specific Aim 3). For the current study, 30 adoptive parent-child dyads (child ages 4-9) will be recruited and randomly assigned to receive one of two interventions. As an inclusion criteria, all children will be required to receive a parent-reported clinically elevated or borderline score on the Total Score of the Strengths and Difficulties Questionnaire (SDQ; ≥ 14) as an index of self-regulation. The SDQ will be used as an outcome measure, as well as a number of other objective report measures, observations, interviews, and child-completed tasks. Dyads will be recruited through the Penn State Children's Hospital's TLC Research and Treatment Center and established partnerships with local adoption agencies.

ELIGIBILITY:
Inclusion Criteria:

* Child is living with an adoptive caregiver
* Caregiver reports a qualifying score for the child on the SDQ
* Fluent in English
* Child is rated by the caregiver with a score of 14 or greater on the full scale of the SDQ.

Exclusion Criteria:

* Child diagnosed with a severe developmental delay and/or psychiatric problem that necessitates a higher level of care.
* IQ below 70 as assessed at the time of the first assessment.

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2019-10-14 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
Strengths and Difficulties Questionnaire (SDQ) | 6 months
  A measure of broadband concerns with emotional, behavioral, cognitive, and social regulation

CONTACTS AND LOCATIONS:
Locations (1):
- Penn State Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No